CLINICAL TRIAL: NCT01929629
Title: A Phase I, Randomized, Placebo-controlled, Single-center Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD0914 After a Single Oral Administration and to Assess the Effect of Food in Healthy Adult Volunteers
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD0914
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D4930C00001
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Gonococcal (GC) Infection
Keywords: Phase 1; Healthy Volunteers; First Time in Man; Pharmacokinetics
MeSH Terms: conditions — Gonorrhea; Infections | interventions — Medicare Part B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo fasting (Placebo Comparator): Single or multiple dosing placebo
  Interventions: Drug: Part A
- Active fed condition (Experimental): AZD0914 given as single dose
  Interventions: Drug: Part B

INTERVENTIONS:
Drug: Part A — Single ascending doses
  Arms: Placebo fasting
Drug: Part B — Single doses food effect. Subjects to receive 2 single doses, one in fed and one in fasted.
  Arms: Active fed condition

SUMMARY:
The purpose of this study is to assess the safety and tolerability of orally administered AZD0914 in healthy adult subjects.

DETAILED DESCRIPTION:
A Phase I, Randomized, Placebo-controlled, Single-center Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD0914 After a Single Oral Administration and to Assess the Effect of Food in Healthy Adult Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (of non-childbearing potential)subjects aged 18 to55 years (inclusive).
* Have a body mass index (BMI) between 18.00 and 30.50 kg/m2 and weigh at least 50 kg and no more than 100 kg
* Male subjects should be willing to use barrier contraception, ie, condoms, from the day of dose administration until at least 3 months after dose administration of the IP

Exclusion Criteria:

* History of any important clinically significant disease or disorder which, in the opinion of the PI, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks from the first administration of IP as judged by the PI
* History of gastrointestinal ulcer disease, inflammatory bowel disease, indigestion symptoms >3 times a week, or blood in stool in previous 6 months not related to anal trauma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Description of the safety profile in terms of adverse events; blood pressure, heart rate and body temperature; electrocardiograms; telemetry; clinical chemistry ; haematology and physical examination | From admission on day -1 until follow up. ( Max 16 days)
  Applies to Part A and B

SECONDARY OUTCOMES:
Description of pharmacokinetics(PK) for AZD0914 study part A and B in terms of maximum observed plasma concentration (Cmax) | Samples taken at predose, and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose
Description of pharmacokinetics(PK) for AZD0914 study part A and B in terms of time to reach maximum observed plasma concentration (tmax) | Samples taken at predose, and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose
Description of pharmacokinetics(PK) for AZD0914(Part A and B) in terms of AUC from time zero to time of last quantifiable AZD0914 concentration [AUC(0-last)] | Samples taken at predose, and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose
Description of pharmacokinetics(PK) for AZD0914(Part A and B) in terms of AUC from time zero to 24 hours after dosing [AUC(0-24)] | Samples taken at predose, and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose
Description of pharmacokinetics(PK) for AZD0914(Part A and B) in terms of terminal half-life (t1/2λz) and apparent plasma clearance (CL/F) | Samples taken at predose, and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose
Description of pharmacokinetics(PK) for AZD0914(Part A and B) in terms of apparent terminal phase volume of distribution (Vz/F), and at steady state (Vss/F),mean residence time | Samples taken at predose, and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose
Description of pharmacokinetics(PK) for AZD0914 (Part A and B) in terms of cumulative amount of investigation product (IP) excreted unchanged into urine from zero to time t [Ae(0-t)], | Samples taken from collections between -12 to 0 hours predose, and 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 48, and 48 to 72 hours after the 1st dose
Description of pharmacokinetics(PK) for AZD0914 (Part A and B) in terms of fraction of dose excreted unchanged into urine (fe), and renal clearance (CLr) | Samples taken from collections between -12 to 0 hours predose, and 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 48, and 48 to 72 hours after the 1st dose

CONTACTS AND LOCATIONS:
Overall Officials: David Mathews, MD, Principal Investigator — Quintiles Phase I unit, Kansas; Humphrey Gardener, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] O'Donnell J, Lawrence K, Vishwanathan K, Hosagrahara V, Mueller JP. Single-Dose Pharmacokinetics, Excretion, and Metabolism of Zoliflodacin, a Novel Spiropyrimidinetrione Antibiotic, in Healthy Volunteers. Antimicrob Agents Chemother. 2018 Dec 21;63(1):e01808-18. doi: 10.1128/AAC.01808-18. Print 2019 Jan. PMID 30373802